CLINICAL TRIAL: NCT01120327
Title: A Pilot Study Exploring Efficacy and Safety of Amlodipine in the Stented Angina Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Hyo-Soo, Kim, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Amlodipine study
Record Dates: First submitted 2010-04-30; First posted 2010-05-10 (Estimated); Last update posted 2010-05-10 (Estimated); Status verified 2010-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Amlodipine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amlodipine (Experimental): Amlodipine
  Interventions: Drug: Amlodipine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Amlodipine — Amlodipine
  Arms: Amlodipine

SUMMARY:
1. OBJECTIVES

   Primary objective to evaluate the difference of the peak oxygen uptake change (VO2 max, mL/kg/min) in amlodipine group against no CCB group at 9 months

   Secondary objectives To evaluate the change of sublingual nitrate use per day against no CCB group at 1 and 3 months To evaluate the change of biomarkers against no CCB group at 9 months
2. SUBJECTS AND CENTERS 212, stable angina patients with angiographically confirmed significant residual stenosis 10, 3rd-grade, teaching hospitals in Korea

ELIGIBILITY:
Inclusion Criteria:

* Stable angina patient with angiographically confirmed significant residual stenosis
* Stenosis more than 50% in 2 major coronary arteries at least or Stenosis more than 75% in 1 major coronary artery

Exclusion Criteria:

* No other pulmonary/psychiatry/musculoskeletal disorder limiting CPET
* Contraindicated to the CPET (e.g. unstable angina, aortic stenosis, uncontrolled hypertension, uncontrolled asthma, hypoxemia at rest, epilepsy, locomotor disorder, severe hypertension and febrile illness)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-07 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | 9 months
  Difference of the peak oxygen uptake change (VO2 max, mL/kg/min)

SECONDARY OUTCOMES:
Sublingual Nitrate | 1month and 3 months
  To evaluate the change of sublingual nitrate use per day against no CCB group at 1 and 3 months
Biomarkers | 9 months
  To evaluate the change of biomarkers against no CCB group at 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea